CLINICAL TRIAL: NCT02384343
Title: Intravenous Dexmedetomidine for Treatment of Shivering During Cesarean Section Under Neuraxial Anesthesia: A Randomized Controlled Trial
Brief Title: Intravenous Dexmedetomidine for Treatment of Shivering During Cesarean Section Under Neuraxial Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Christina Lamontagne, MD, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 050115
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Tremor
Keywords: Dexmedetomidine; Cesarean section; Anesthesia, Spinal; Anesthesia, Epidural
MeSH Terms: conditions — Tremor | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine 4 mcg/ml, 30 mcg (7,5 ml), single intravenous bolus
  Interventions: Drug: Dexmedetomidine
- Normal saline (Placebo Comparator): NaCl 0,9% 7,5 ml, single intravenous bolus
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — An intravenous bolus of dexmedetomidine 30 mcg (7,5 mL) administered at least five minutes after birth, in participants with shivering grade 3 or 4 on a scale described by Crossley and Mahajan.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Normal saline — An intravenous bolus of normal saline (7,5 mL) administered at least five minutes after birth, in participants with shivering grade 3 or 4 on a scale described by Crossley and Mahajan.
  Other Names: NaCl 0,9%
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine whether dexmedotomidine is effective in the treatment of shivering associated with neuraxial anesthesia during cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery under neuraxial anesthesia (epidural or spinal) planned or unplanned between 8 am and 8 pm on week days when one of the investigator is present.
* Participants with fever or shivering before the cesarean section are include

Exclusion Criteria:

* No comprehension of french or english language
* Urgent cesarean delivery for non reassuring fetal tracing
* Extremely urgent cesarean delivery (grade 1)
* Weight < 60 kg ou > 120 kg
* Hypersensibility to dexmedetomidine
* Heart, renal or hepatic disease requiring follow up, medication or with a possibility of instability during cesarean delivery
* Pre-eclampsia
* Combined spinal-epidural anesthesia
* Conversion into general anesthesia
* Blood products transfusions or major complications during surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Time for cessation of shivering after bolus (min) | Within the first 15 minutes of administration of bolus
  Graded on a four point scale as per Crossley and Mahajan

SECONDARY OUTCOMES:
Incidence of bradycardia | From the administration of bolus to the end of surgery, an expected average of 1 hour
  Heart rate below 50 bpm
Incidence of hypotension | From the administration of bolus to the end of surgery, an expected average of 1 hour
  A decrease in mean arterial pressure by more than 20% of the baseline mean arterial pressure
Incidence of sedation | From the administration of bolus to the end of surgery, an expected average of 1 hour
  Graded on a four point scale as per Filos et al

CONTACTS AND LOCATIONS:
Overall Officials: Christina Lamontagne, MD, Principal Investigator — St. Justine's Hospital; Chantal Crochetière, MD, FRCP, Study Director — St. Justine's Hospital; Edith Villeneuve, Study Chair — St. Justine's Hospital; Sandra Lesage, Study Chair — St. Justine's Hospital
Locations (1):
- St-Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mittal G, Gupta K, Katyal S, Kaushal S. Randomised double-blind comparative study of dexmedetomidine and tramadol for post-spinal anaesthesia shivering. Indian J Anaesth. 2014 May;58(3):257-62. doi: 10.4103/0019-5049.135031. PMID 25024466
- [Background] Crowley LJ, Buggy DJ. Shivering and neuraxial anesthesia. Reg Anesth Pain Med. 2008 May-Jun;33(3):241-52. doi: 10.1016/j.rapm.2007.11.006. PMID 18433676
- [Background] Crossley AW, Mahajan RP. The intensity of postoperative shivering is unrelated to axillary temperature. Anaesthesia. 1994 Mar;49(3):205-7. doi: 10.1111/j.1365-2044.1994.tb03422.x. PMID 8147511
- [Derived] Lamontagne C, Lesage S, Villeneuve E, Lidzborski E, Derstenfeld A, Crochetiere C. Intravenous dexmedetomidine for the treatment of shivering during Cesarean delivery under neuraxial anesthesia: a randomized-controlled trial. Can J Anaesth. 2019 Jul;66(7):762-771. doi: 10.1007/s12630-019-01354-3. Epub 2019 Apr 3. PMID 30945105